CLINICAL TRIAL: NCT06430008
Title: A Study to Explore the Correlation Between Total Sialic Acid Combined With Superoxide Dismutase and the Diagnosis and Prognosis of Lipoid Pneumonia
Brief Title: The Relationship Between Total Sialic Acid and Superoxide Dismutase and the Diagnosis and Prognosis of Lipoid Pneumonia
Status: Enrolling by invitation | Type: Observational
Sponsor: Hu Yinan (Other)
Responsible Party: Sponsor-Investigator, Hu Yinan, China-Japan Friendship Hospital, China-Japan Friendship Hospital
Organization: China-Japan Friendship Hospital (Other)
Other Study IDs: 2024-KY-144
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Lipid Pneumonia; Superoxide Dismutase; Sialic Acid
MeSH Terms: conditions — Pneumonia, Lipid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- lipid pneumonia
- cough
- cryptogenic organizing pneumonia
- pulmonary alveolar proteinosis
- bacterial pneumonia
- fungal pneumonia
- pulmonary edema
- mucinous adenocarcinoma of the lung

SUMMARY:
The goal of this observational study is to explore the correlation between total sialic acid combined with superoxide dismutase and the diagnosis and prognosis of lipid pneumonia in the patient with lipid pneumonia, cough, bacterial and fungal pneumonia, cryptogenic organizing pneumonia, pulmonary alveolar proteinosis, lung mucinous adenocarcinoma and pulmonary edema. The main question it aims to answer is:

Whether superoxide dismutase (SOD) and total sialic acid (TSA) could be used as diagnostic markers to distinguish lipid pneumonia from patient with cough, and bacterial and fungal pneumonia, cryptogenic organizing pneumonia, pulmonary alveolar proteinosis, lung mucinous adenocarcinoma and pulmonary edema, whether SOD and TSA be associated with the prognosis of patients with lipid pneumonia?

Participants will answer online survey questions about their symptoms, changes in oxygen status, and changes in the most recent CT image of the lung for up to 10 years after treatment. We will count participants' baseline data including: gender, age, smoking history, comorbidities, lung function, imaging findings, hormone use or not, ICU treatment, death or not, the type of cause of lipid pneumonia, how it is diagnosed, and their baseline SOD and TSA.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥ 18 years old;
2. The diagnosis of lipoid pneumonia must be supported by lung biopsy pathological support or positive oil red O or Sudan staining in bronchoalveolar lavage fluid;
3. Patients with bacterial and fungal pneumonia must be supported by etiological evidence;
4. Patients with cryptogenic organizing pneumonia and pulmonary alveolar proteinosis must be supported by lung biopsy pathology;
5. Patients with lung mucinous adenocarcinoma must be supported by lung tissue biopsy;
6. Lung imaging of patients with pulmonary edema must show paving stone signs;

Exclusion Criteria:

1. Age< 18 years old;
2. The patient only has a history of lipid inhalation and no pathology or positive lipoid staining;
3. Co-infection with the corona virus disease 2019 at the onset of illness;
4. Pregnant

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study includes the lipoid pneumonia patients, patients with cough in the upper respiratory tract only, patients with bacterial and fungal pneumonia, patients with cryptogenic organizing pneumonia and pulmonary alveolar proteinosis, patients with lung mucinous adenocarcinoma and patients with pulmonary edema.
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
superoxide dismutase | At the time of admission

SECONDARY OUTCOMES:
sialic acid | At the time of admission
death or not | Within 10 years after discharge
neutrophil-to-lymphocyte ratio | At the time of admission

CONTACTS AND LOCATIONS:
Overall Officials: Yinan Hu, Study Chair — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected throughout the trial, only IPD used in the results publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
URL: http://www.medresman.org.cn

REFERENCES:
- [Derived] Hu Y, Ren Y, Han Y, Li Z, Meng W, Qiang Y, Liu M, Dai H. Relevance of superoxide dismutase type 1 to lipoid pneumonia: the first retrospective case-control study. Respir Res. 2025 Jan 18;26(1):24. doi: 10.1186/s12931-025-03101-3. PMID 39827104